CLINICAL TRIAL: NCT00652639
Title: Comparative, Randomized, Single-Dose, 2 Way Cross Over Bioavailability Study of Kali's Clonazepam Tablets 1 mg With That of Klonopin Tablets 1 mg in Healthy Adult Subjects Under Fasting Conditions.
Brief Title: Bioavailability Study of Clonazepam Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Cetero Research, San Antonio (Network)
Responsible Party: Dr. Alfred Elvin/ Director Biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B043201
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-04

CONDITIONS: To Determine Bioequivalence Under Fasting Conditions
Keywords: bioequivalence, Clonazepam tablets, fasting
MeSH Terms: conditions — Fasting | interventions — Clonazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received the kali formulated products under fasting conditions
  Interventions: Drug: Clonazepam
- B (Active Comparator): Subjects received the Roche formulated products under fasting conditions
  Interventions: Drug: Klonopin

INTERVENTIONS:
Drug: Clonazepam — Tablets, 1 mg, single-dose
  Other Names: Klonopin
  Arms: A
Drug: Klonopin — tablets, 1 mg, single-dose
  Other Names: Clonazepam tablets
  Arms: B

SUMMARY:
To compare the single-dose bioavailability of Clonazepam tablets 1 mg and Klonopin tablets 1 mg

DETAILED DESCRIPTION:
To compare the single -dose bioavailability of kali's Clonazepam tablets 1 mg with that of Klonopin tablets 1 mg by Roche pharmaceuticals following a single oral dose under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* All subjects selected for this study will be alt least 18 years of age.Females must be of non- childbearing potential (postmenopausal for alt least 6 months or surgically sterile)
* Each subject shall be given a general physical examination within 28 days of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history.
* Each female subject will be given a serum pregnancy test as part of the pre-study process.
* At the end of the study, the subjects will have an exit evaluation consisting of interim history, global evaluation, and clinical laboratory measurements.
* Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trail for clinical laboratory.
* Clinical laboratory measurements will include the following:
* Hematology: hemoglobin, hematocrit, red blood cell count (with differential)
* Clinical Chemistry: creatinine, BUN, glucose, SGOT/ AST, SGPT/ALT, bilirubin, and alkaline phosphate.
* Urine Analysis: pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood and cells.
* HIV Screen: (Pre-study only)
* Hepatitis-B, C Screen: (Pre-study only)
* Drugs of Abuse Screen: (Pre-study at check -in each dosing period)
* Electrocardiograms of all participating subjects will be recorded before initiation of the study and filed with each subject's case report forms.

Exclusion Criteria:

* Subjects with a history of chronic alcohol consumption (during past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis epilepsy, asthma, (during pat 5 years), diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are outside the normal range may be retested at the discretion of the clinical investigator. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
* Subjects who have a history of allergic response to the class of drug being tested should excluded form the study.
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and check in each dosing period. Subjects found to have urine concentration of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/plasma for at least thirty (30) days prior to the first dosing of the study
* Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Female subjects with childbearing potential will not be allowed to participate.
* All female subjects will be screened for pregnancy at check in each study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-02; Primary Completion 2004-03 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Plisco, Principal Investigator — Cetero Research, San Antonio; Gary Shillito, Study Director — Cetero Research, San Antonio